CLINICAL TRIAL: NCT00378378
Title: Study of Nasonex® for the Treatment of Nasal Polyps in Pediatric Subjects Between Ages of 6 and Less Than 18 Years Old
Brief Title: Study of Nasonex® for the Treatment of Nasal Polyps in Pediatric Subjects Between Ages of 6 and Less Than 18 Years Old (P04292)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04292
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- MFNS 100 mcg QD for subjects 6 to less than 12 years (Experimental): Mometasone Furoate nasal Spray (MFNS) 100 mcg once per day (QD) for subjects 6 to less than 12 years of age
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)
- Placebo QD for subjects 6 to less than 12 years (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray
- MFNS 200 mcg QD for subjects 12 to less than 18 years (Experimental)
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)
- MFNS 200 mcg BID for subjects 12 to less than 18 years (Experimental)
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)
- Placebo QD for subjects 12 to less than 18 years (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray
- MFNS 100 mcg BID for subjects 6 to less than 12 years (Experimental)
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)
- Placebo BID for subjects 6 to less than 12 years (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray
- Placebo BID for subjects 12 to less than 18 years (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray (MFNS) — 100 mcg nasal spray
  Other Names: Nasonex
  Arms: MFNS 100 mcg BID for subjects 6 to less than 12 years; MFNS 100 mcg QD for subjects 6 to less than 12 years; MFNS 200 mcg BID for subjects 12 to less than 18 years; MFNS 200 mcg QD for subjects 12 to less than 18 years
Drug: Placebo nasal spray — One spray of placebo nasal spray in each nostril once daily for 4 months.
  Arms: Placebo BID for subjects 12 to less than 18 years; Placebo BID for subjects 6 to less than 12 years; Placebo QD for subjects 12 to less than 18 years; Placebo QD for subjects 6 to less than 12 years

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Nasonex® (Mometasone Furoate Nasal Spray(MFNS)) in the treatment of nasal polyps in pediatric subjects between the ages of 6 and less than 18 years old. Safety will be the primary focus of this study.

ELIGIBILITY:
Inclusion Criteria:

* A subject must be 6 to <18 years of age, of either sex, and of any race.
* A subject must have a diagnosis of bilateral nasal polyps.
* A subject must have a minimum nasal congestion/obstruction
* An asthmatic subject may be included.
* A subject's clinical laboratory tests (hematology, blood chemistry, and urinalysis) must be within normal limits or clinically acceptable to the investigator/sponsor.
* The subject and parent/guardian must be willing to give written informed consent, and the subject must be able to adhere to dose and visit schedules.
* A female subject of child-bearing potential who is sexually active must have been using a medically accepted method of contraception prior to Screening and must continue using it while receiving protocol-specified medication. If a pre-menarche female subject begins menstruating during the study, a serum pregnancy test must be done at the next visit

Exclusion Criteria:

* A subject with antrochoanal polyps.
* A subject with cystic fibrosis.
* A subject with acute sinusitis, concurrent upper respiratory tract infection, or who had an upper respiratory tract infection within 2 weeks prior to the Screening Visit.
* A subject with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
* A subject who is immunocompromised.
* A subject with ongoing rhinitis medicamentosa.
* A subject with Churg Strauss syndrome.
* A subject with dyskinetic ciliary syndromes, eg, Young's syndrome (sinopulmonary infections and obstructive azoospermia) or Kartagener's syndrome (immotile cilia).
* A subject with any clinically significant pretreatment laboratory, vital sign, or ECG abnormality.
* A subject with allergy/sensitivity to aspirin, corticosteroids, or study drug or its excipients.
* A subject who has not observed the medication washout times outlined in the protocol prior to the Screening Visit.
* A female subject who is breast-feeding, pregnant, or intends to become pregnant.
* A subject who has used any investigational drug within 30 days of Screening.
* A subject who is part of the staff personnel directly involved with this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chur V, Small CB, Stryszak P, Teper A. Safety of mometasone furoate nasal spray in the treatment of nasal polyps in children. Pediatr Allergy Immunol. 2013 Feb;24(1):33-8. doi: 10.1111/pai.12032. PMID 23331528

RESULTS

PARTICIPANT FLOW:
Groups:
- MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years: Subjects 6 to less than 12 years of age were pooled for Mometasone Furoate Nasal Spray (MFNS) twice per day (BID)
- MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years: Subject 12 to less than 18 years of age were pooled for Mometasone Furoate Nasal Spray (MFNS) once per day (QD)
- Pooled Placebo: All placebo groups were combined
Period: Overall Study
Arm/Group | MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years | MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years | Pooled Placebo
Started | 51 | 50 | 26
Completed | 51 | 49 | 24
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Treatment Failure | 0 | 0 | 1
Not completed — Non-compliance with protocol | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years | MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years | Pooled Placebo | Total
Number analyzed (Participants) | 51 | 50 | 26 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.4) | 14.4 (1.8) | 12.7 (3.2) | 12.7 (2.9)
Age, Customized [Number; unit: participants]
  6 to < 12 years | 18 | 18 | 10 | 46
  12 to < 18 years | 33 | 32 | 16 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 12 | 54
  Male | 31 | 28 | 14 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline 24-hour Urinary Free Cortisol Level
Description: The primary objective of this study was to evaluate the safety of Mometasone Furoate Nasal Spray (MFNS) in the treatment of pediatric subjects 6 to <18 years of age. Primary safety was to be assessed by determining the subject's 24-hour urinary free cortisol level.
Time Frame: Baseline to Endpoint
Population: Not all participants that were randomized had both a baseline and an endpoint urine sample. Only participants with both were included in the participants analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mcg/hour
Arm/Group | MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years | MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years | Pooled Placebo
Number analyzed (Participants) | 44 | 50 | 25
mcg/hour
  Baseline | 49.5 (32.4) | 39.6 (32.4) | 49.8 (32.4)
  Change from Baseline to Endpoint | 1.5 (42.9) | 11.6 (42.9) | -2.1 (42.9)
Statistical Analysis 1: Comparison: MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years vs MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years; Pairwise comparison p-values were based on a two-way ANOVA for the change from basline; Test type: Superiority or Other; p = 0.258, ANOVA
Statistical Analysis 2: Comparison: MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years vs Pooled Placebo; Pairwise comparison p-values were based on a two-way ANOVA for the change from baseline; Test type: Superiority or Other; p = 0.735, ANOVA
Statistical Analysis 3: Comparison: MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years vs Pooled Placebo; Pairwise comparison p-values were based on a two-way ANOVA for the change from baseline; Test type: Superiority or Other; p = 0.194, ANOVA

2. Secondary Outcome: Change From Baseline 24-hour Urinary Free Cortisol Level Corrected for Creatinine
Description: The key secondary objective of this study was the assessment of the 24-hour urinary free cortisol level (corrected for creatinine).
Time Frame: Baseline to Endpoint
Measure: Least Squares Mean (Standard Deviation); unit: mcg/hour
Arm/Group | MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years | MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years | Pooled Placebo
Number analyzed (Participants) | 44 | 50 | 25
mcg/hour
  Baseline | 6.7 (4.5) | 5.3 (4.5) | 7.6 (4.5)
  Baseline to Endpoint | 0.0 (4.9) | 1.0 (4.9) | -0.6 (4.9)
Statistical Analysis 1: Comparison: MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years vs MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years; Pairwise comparison p-values were based on a two-way ANOVA for baseline to endpoint; Test type: Superiority or Other; p = 0.361, ANOVA
Statistical Analysis 2: Comparison: MFNS 100 or 200 mcg BID for Subjects 6 to Less Than 18 Years vs Pooled Placebo; Pairwise comparison p-values were based on a two-way ANOVA for baseline to endpoint; Test type: Superiority or Other; p = 0.603, ANOVA
Statistical Analysis 3: Comparison: MFNS 100 or 200 mcg QD for Subjects 6 to Less Than 18 Years vs Pooled Placebo; Pairwise comparison p-values were based on a two-way ANOVA for baseline to endpoint; Test type: Superiority or Other; p = 0.193, ANOVA

ADVERSE EVENTS:
Arm/Group | MFNS 100 or 200 mcg QD | MFNS 100 or 200 mcg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/26
Other Adverse Events (participants affected / at risk) | 24/50 | 23/51 | 13/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS 100 or 200 mcg QD (N=50) | MFNS 100 or 200 mcg BID (N=51) | Placebo (N=26)
EAR PAIN (Ear and labyrinth disorders) | 3 (6) | 1 (4) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 3 (3) | 1 (2)
INFLUENZA (Infections and infestations) | 4 (4) | 4 (6) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 6 (6) | 6 (8)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (4) | 2 (2)
HEADACHE (Nervous system disorders) | 12 (32) | 10 (22) | 8 (14)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 6 (32) | 1 (3)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 1 (2) | 1 (3)

LIMITATIONS AND CAVEATS:
The standard deviation is pooled for Primary and Secondary Outcome Measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less